A single-blind, parallel-group randomised trial of a Technology-assisted and remotely delivered Cognitive Behavioural Therapy intervention (Tech-CBT) versus usual care to reduce anxiety in people with mild cognitive impairment and dementia:

# Statistical Analysis Plan

Version 1.0, Dated 29 January 2026

The preparation of this document has been led by the trial statistician, who will remain blinded until this document has been agreed and uploaded to: <a href="https://clinicaltrials.gov/study/NCT05528302">https://clinicaltrials.gov/study/NCT05528302</a>.

This document has been approved by the following:

| Position | Name |
|------------------------|--------------------------|
| Principal Investigator | Prof Nadeeka Dissanayaka |
| Trial statistician | Mark Chatfield |
| Investigator | Adam Charters |
| Investigator | Dr Deborah Brooks |
| Investigator | Dr Leander Mitchell |
| Investigator | Tiffany Au |

## Introduction

The study protocol has been published in *Trials*: <a href="https://doi.org/10.1186/s13063-023-07381-2">https://doi.org/10.1186/s13063-023-07381-2</a>

This document describes how the quantitative data (with the exception of the health economic data) will be reported and analysed in the main results publication.

# Reporting and analysis of outcomes

In the protocol (and on the trial registry), one primary outcome and 11 secondary outcomes were listed. Some detail on the outcome measures is provided in the Table below. The primary timepoint is T2 (Week 8).

Table. Outcomes

| | | Range | Baseline | | Post-baseline | |
|---|---|---|---|---|---|---|
| | | | T1 | T2 (Week 8) | T3 (Week 20) | T4 (Week 32) |
| | Primary Outcome | | | | | |
| | Rating Anxiety in Dementia (RAID) | 0 - 54 | X | Х | Х | X |
| | Secondary Outcomes | | | | | |
| | -All participants living with MCI/dementia- | | | | | |
| 1 | Quality of life in Alzheimer's disease (QoL-AD) | <b>13</b> – 52 | X | Х | Х | Х |
| 2 | Geriatric Anxiety Inventory (GAI) | 0 - 20 | X | Х | Х | Х |
| 3 | Penn State Worry Questionnaire (PSWQ-A) | 8 - 40 | X | Х | Х | Х |
| 4 | Perceived Stress Scale (PSS-14) | 0 - 56 | X | Х | Х | Х |
| 5 | Geriatric Depression Scale (GDS-15) | 0 - 15 | X | Х | Х | X |
| | -People living with PD and MCI/dementia- | | | | | |
| 6 | Parkinson's Anxiety Scale (PAS) | 0 - 48 | X | Χ | | |
| 7 | Parkinson's disease Specific Anxiety Inventory (PDSAI) | 0 - 40 | Х | Χ | | |
| 8 | Patient Reported Outcomes in Parkinson's Disease (PRO-PD) | 0 - 3500 | X | Х | X | Х |
| | -Support persons- | | | | | |
| 9 | Zarit Burden Inventory (ZBI) | 0 - 88 | Х | Χ | X | X |
| 10 | Assessment of quality of life (AQoL-6D) | 20 - 99 | X | Χ | Х | X |
| 11 | Depression, Anxiety and Stress Scale (DASS-21) | 0 - 126 | X | Χ | | |

Note. Worst score coloured in red.

#### Analysis of primary outcome and secondary outcomes 1-5 and 9-10

We will use a linear mixed model to estimate adjusted between-group differences in change from baseline at the post-baseline timepoints. The model will include fixed effects for the outcome at baseline, gender of participant living with MCI/dementia, randomisation group, post-baseline timepoint (i.e. T2, T3 or T4) and interactions between group and timepoint. Participant will be a random effect. The model will be fit via restricted maximum likelihood (REML) and the Kenward-Roger method used for computing degrees of freedom of a t-distribution.

i.e.
on a dataset that looks like this:

| 1001 | tcome | change_out | baseline | outcome | time | randgroup | record_id |
|---|---|---|---|---|---|---|---|
| 1001 2 3 5 28 | -19 | | 28 | 9 | 2 | 2 | 1001 |
| | -23 | | 28 | 5 | 3 | 2 | 1001 |
| 1001 2 4 14 28 | -14 | | 28 | 14 | 4 | 2 | 1001 |

the following Stata syntax will be used to estimate the between-group difference (intervention(1) – control(2)) in change from baseline

at T2: . mixed change\_outcome baseline ib2.randgroup##ib2.time i.gender if time>1 || record\_id:, reml dfmethod(kroger)

at T3: . mixed change\_outcome baseline ib2.randgroup##ib3.time i.gender if time>1 || record\_id:, reml dfmethod(kroger)

at T4: . mixed change\_outcome baseline ib2.randgroup##ib4.time i.gender if time>1 || record\_id:, reml dfmethod(kroger)

Note, the above syntax fits the same model (three times). It just expresses the model in different ways, so that the between-group differences at T2, T3 and T4 can be obtained with the Kenward-Roger DF method.

#### Analysis of secondary outcome 11 (DASS, just assessed at T1 and T2)

We will use an ANCOVA model to estimate the between-group difference in change from baseline at T2. Fixed effects will be randomisation group, gender of the participant living with MCI/dementia and the outcome at baseline.

The following Stata syntax will be used:

. regress change\_outcome baseline ib2.randgroup i.gender if time==2

#### Analysis of secondary outcomes 6-8

Due to limited post-baseline data\*, there will be no analysis of the outcomes for participants living with PD and MCI/dementia.

\*At a post-baseline timepoint, no more than n=3 will have data for one of these outcomes.

#### Presenting data and analyses

We will report the data relating to the outcomes in the tables below,

and produce line graphs showing mean outcome and 95%CI for each group at each timepoint, calculated using syntax like this:

- . mixed outcome time#randgroup i.gender || record\_id:, reml
- . margins time#randgroup
- . marginsplot

**Table 1**Baseline Characteristics, by Randomised Group

| Variable | Tech-CBT | Group ( <i>n</i> = ) | TAU Gr | oup (n = ) | _ Test Statistic |
|---|---|---|---|---|---|
| variable | n (%) | Mean (SD) | n (%) | Mean (SD) | _ Test Statistic |
| Age | | | | | |
| Gender (% female) | | | | | |
| Diagnostic aetiology | | | | | |
| MCI | | | | | _ |
| Dementia | | | | | _ |
| TICS-M | | | | | |
| IADL | | | | | |
| Participating with support person | | | | | |
| Language other than English | | | | | |
| Living in regional or remote area <sup>a</sup> | | | | | |
| Years of formal education | | | | | |
| Subjective reports of anxiety | | | | | |
| Self-report diagnosis of anxiety disorder | | | | | _ |
| Self-report diagnosis of depressive disorder | | | | | _ |

Note. N people living with cognitive impairment = . n = 1 support person did not provide baseline responses. TAU = Treatment as usual. SD = Standard deviation. MCI = Mild Cognitive Impairment. TICS-M = Modified Telephone Interview for Cognitive Status. IADL = Lawton Instrumental Activities of Daily Living. Test statistic is t(df) for continuous data and  $\chi^2(1)$  for categorical data.

<sup>&</sup>lt;sup>a</sup> Rural or Regional area defined as Modified Monash Model classification 2-7 (2023).

\*p < .05, \*\*p < .01, \*\*\*p < .001

Figure 1

CONSORT Flowchart of Screened Participants



*Note. TAU* = Treatment as usual. StepUp for Dementia Research is funded by the Australian Government Department of Health and implemented by a dedicated team at the University of Sydney (Jeon et al., 2021).

 Table 2

 Outcomes for People Living with Cognitive Impairment and their Support Persons

| | | | | | Post | 3-Month | 6-Month |
|---|---|---|---|---|---|---|---|
| | Baseline M(SD) | Post M(SD) | 3-Month M(SD) | 6-Month M(SD) | adjusted mean | adjusted mean | Adjusted mean |
| | | | | | difference | difference | difference |
| | | | | | (95% CI) | (95% CI) | (95% CI) |
| | | Measure | es for People Living with | Cognitive Impairment | | | |
| RAID | | | | | | | |
| Tech-CBT | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x [x.x, x.x]* | x.x [x.x, x.x]* | x.x [x.x, x.x]* |
| TAU | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | | | |
| GAI | | | | | | | |
| Tech-CBT | | | | | | | |
| TAU | | | | | | | |
| PSWQ-A | | | | | | | |
| Tech-CBT | | | | | | | |
| TAU | | | | | | | |
| PSS-14 | | | | | | | |
| Tech-CBT | | | | | | | |
| TAU | | | | | | | |
| GDS-15 | | | | | | | |
| Tech-CBT | | | | | | | |
| TAU | | | | | | | |
| QoL-AD | | | | | | | |
| Tech-CBT | | | | | | | |

#### Measures for Support Persons

AQoL

Tech-CBT

TAU

ZBI

Tech-CBT

TAU

DASS-21

Tech-CBT

TAU

Note. M = Mean. SD = Standard deviation. RAID = Rating Anxiety in Dementia. TAU = Treatment as usual. GAI = Geriatric Anxiety Inventory. PSWQ-A = Penn State Worry

Questionnaire. GDS-15 = Geriatric Depression Scale. QoL-AD = Quality of Life in Alzheimer's Disease. AQoL = Assessment of Quality of Life. ZBI = Zarit Burden Inventory.

DASS-21 = Depression, Anxiety and Stress Scale 21.

\**p* < .05. \*\**p* < .01. \*\*\**p* < .001.

Figure 2

Rating Anxiety in Dementia Mean Scores at Each Timepoint



*Note.* For readability, line graphs showing the mean and 95% confidence interval of each outcome will be provided in the supplementary of the article, unless a notable trend emerges that warrants discussion in the main text.

Supplementary Table 1

More information on Outcomes for People Living with Cognitive Impairment and their Support Persons

| Outcome | Timepoint | Group | n | Mean (SD) | Between-<br>group $t(df)^a$ | <i>n</i> change | Mean change<br>(SD) | Adjusted mean difference (95% CI) |
|---|---|---|---|---|---|---|---|---|
| | | | Measures for P | eople Living with Co | gnitive Impairment | | | |
| | Baseline | Tech-CBT | Х | Х | X* | | | |
| | ваѕеппе | TAU | Х | X | | | | |
| | Doct | Tech-CBT | Х | X | | Χ | X | X [X , X]* |
| 2412 | Post | TAU | Х | X | | Χ | X | |
| RAID | 3-Month | Tech-CBT | Х | X | | X | X | X [X , X]* |
| | | TAU | Х | X | | X | X | |
| | 6-Month | Tech-CBT | Х | X | | X | X | X [X , X]* |
| | | TAU | Х | X | | Χ | X | |
| | Baseline | Tech-CBT | | | | | | |
| | | TAU | | | | | | |
| | | Tech-CBT | | | | | | |
| CAL | Post | TAU | | | | | | |
| GAI | 2.84 | Tech-CBT | | | | | | |
| | 3-Month | TAU | | | | | | |
| | C NA south | Tech-CBT | | | | | | |
| | 6-Month | TAU | | | | | | |
| DCM/O A | Deseline | Tech-CBT | | | | | | |
| PSWQ-A | Baseline | TAU | | | | | | |

| Fost | | Doct | Tech-CBT |
|---|---|---|---|
| 3-Month | | FOST | TAU |
| TAU Tech-CBT TAU Baseline TECH-CBT TAU Post TAU Post TAU 3-Month TAU Tech-CBT TAU TAU Tech-CBT TAU TAU Tech-CBT TAU TAU Tech-CBT TAU TAU TAU TAU TECH-CBT TAU TAU TAU TECH-CBT TAU TAU TAU TECH-CBT TAU TAU TECH-CBT TAU TAU TECH-CBT TECH-CBT | | 3-Month | Tech-CBT |
| Factor F | | | TAU |
| TAU | | C. N. A. o. o. t. b. | Tech-CBT |
| Baseline TAU Post TECh-CBT 3-Month TECh-CBT TECh-CBT TECh-CBT TAU TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT TECh-CBT <tr< td=""><td></td><td>6-Month</td><td>TAU</td><td></td><td></td></tr<> | | 6-Month | TAU |
| TAU Post Tech-CBT TAU PSS-14 PSS-14 TECH-CBT 3-Month TAU TECH-CBT TAU TECH-CBT TAU TECH-CBT TAU TAU TECH-CBT TAU TAU TECH-CBT TAU | | Deceline | Tech-CBT |
| PSS-14 TAU Tech-CBT 3-Month TAU Tech-CBT | | Baseiine | TAU |
| PSS-14 TECh-CBT 3-Month TAU Tech-CBT TAU Tech-CBT TAU Tech-CBT TAU Post Tau Tech-CBT TAU Tech-CBT | | Doct | Tech-CBT |
| Tech-CBT TAU TAU Tech-CBT TAU TAU Tech-CBT TAU TAU Tech-CBT TAU TAU TEch-CBT TAU TAU TEch-CBT TAU TEch-CBT TAU TEch-CBT TAU Tech-CBT TAU Tech-CBT TAU | DCC 14 | POST | TAU |
| TAU Tech-CBT TAU 6-Month TAU Tech-CBT TAU | P33-14 | 2 Month | Tech-CBT |
| GDS-15 GDS-15 GDS-15 Tech-CBT Tau Tech-CBT | | 3-101011111 | TAU |
| TAU Tech-CBT | | C. N. A. o. o. t. b. | Tech-CBT |
| Baseline TAU Post Tech-CBT TAU Tech-CBT 3-Month TAU Tech-CBT TAU Tech-CBT TAU Tech-CBT TAU Tech-CBT TAU Tech-CBT TAU Au Tech-CBT Tau Tech-CBT | | 6-Month | TAU |
| TAU Tech-CBT Post TAU Tau Tech-CBT 3-Month TAU Tech-CBT Tech-CBT Tau Tech-CBT Tau Tech-CBT Tau Tech-CBT Tau Tech-CBT Tau Tech-CBT | | Pacalina | Tech-CBT |
| GDS-15 TAU Tech-CBT 3-Month TAU Tech-CBT TAU Tech-CBT TAU Tech-CBT TAU Tech-CBT TAU Tech-CBT | | Daseille | TAU |
| GDS-15 Tech-CBT 3-Month TAU Tech-CBT Tau Tech-CBT TAU Tech-CBT TAU TAU Tau Tech-CBT Tau Tech-CBT | | Post | Tech-CBT |
| $\begin{array}{c} \text{Tech-CBT} \\ \text{TAU} \\ \text{6-Month} \end{array}$ $\begin{array}{c} \text{Tech-CBT} \\ \text{TAU} \\ \text{TAU} \\ \\ \text{QoL-AD} \end{array}$ $\begin{array}{c} \text{Baseline} \end{array}$ | GDS-15 | POSI | TAU |
| | GD3-13 | 2-Month | Tech-CBT |
| 6-Month TAU Tech-CBT QoL-AD Baseline | | 3-WOULT | TAU |
| TAU Tech-CBT QoL-AD Baseline | | 6-Month | Tech-CBT |
| QoL-AD Baseline | | o Wollen | TAU |
| TAU | Ool-AD | Baseline | Tech-CBT |
| | QUETID | Baseline | TAU |

| | Post | Tech-CBT | |
|---------|-------------|----------|------------------------------|
| | FOST | TAU | |
| | 3-Month | Tech-CBT | |
| | 3-1011111 | TAU | |
| | 6-Month | Tech-CBT | |
| | 0-IVIOIILII | TAU | |
| - | | | Measures for Support Persons |
| - | Baseline | Tech-CBT | |
| DASS-21 | baseiiile | TAU | |
| DA33-21 | Post | Tech-CBT | |
| | FOSI | TAU | |
| | Baseline | Tech-CBT | |
| | baseine | TAU | |
| | Post | Tech-CBT | |
| ZBI | FOST | TAU | |
| ZDI | 3-Month | Tech-CBT | |
| | 3-101011111 | TAU | |
| | 6-Month | Tech-CBT | |
| | 0-IVIOTICIT | TAU | |
| | Baseline | Tech-CBT | |
| | Daseille | TAU | |
| AQoL | Post | Tech-CBT | |
| | PUSI | TAU | |
| | 3-Month | Tech-CBT | |

TAU

6-Month

Tech-CBT

TAU

Note. SD = Standard deviation. RAID = Rating Anxiety in Dementia. TAU = Treatment as usual. GAI = Geriatric Anxiety Inventory. PSQQ-A = Penn State Worry Questionnaire.

GDS-15 = Geriatric Depression Scale. QoL-AD = Quality of Life in Alzheimer's Disease. AQoL = Assessment of Quality of Life. ZBI = Zarit Burden Inventory. DASS-21 = Depression, Anxiety and Stress Scale 21.

<sup>&</sup>lt;sup>a</sup> Between-group *t*(df) refers to differences between groups at baseline.

### **Supplementary Table 3**

### Differences Between Completers and Non-Completers

| Characteristic | Completed RAID post-assessment | Did not complete RAID post-assessment | Test Statistic |
|---|---|---|---|
| | (n = ) | (n = ) | |
| | Sociodemograp | hic Characteristics | |
| Age | | | |
| Gender (% female) | | | |
| Diagnostic aetiology | | | |
| MCI | | | _ |
| Dementia | | | _ |
| Participating with support person | | | |
| Language other than English | | | |
| Living in regional or remote area | | | |
| Years of formal education | | | |
| Subjective reports of anxiety | | | |
| Self-report diagnosis of anxiety disorder | | | _ |
| Self-report diagnosis of depressive | | | _ |
| disorder | | | |
| | Baseline | e Measures | |
| RAID | | | |
| GAI | | | |
| PSWQ-A | | | |
| PSS-14 | | | |
| GDS-15 | | | |

TICS-M

IADL

QoL-AD

ZBI

AQoL

DASS-21

#### Missing data

When a whole questionnaire/scale is missing at T1/T2/T3/T4, we will NOT impute a total/score.

Therefore, in order to include a person's data in an analysis of an outcome, we need the person to have i) the outcome at baseline and ii) at least one outcome post-baseline.

When just one item is missing from a questionnaire/scale, a total will be calculated by utilising their item score from the most recent administration.